CLINICAL TRIAL: NCT04768140
Title: The Effect Of Bobath Approach On Hemiplegic Shoulder Pain, Spasticity And Upper Extremity Functionality In Stroke Patients: A Prospective, Randomized, Controlled And Single-Blind Trial
Brief Title: Bobath Approach On Hemiplegic Shoulder Pain
Acronym: BAHSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, NAZLI GÜNGÖR, Research Assistant, Department of Physiotherapy and Rehabilitation, Health Sciences School, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAHSP
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: Hemiplegia; hemiplegic shoulder pain; neurodevelopmental treatment; spasticity; stroke
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity; Stroke

STUDY DESIGN:
Intervention Model Description: A PROSPECTIVE, RANDOMIZED, CONTROLLED AND SINGLE-BLIND TRIAL
Who Masked: Participant
Masking Description: SINGLE-BLIND TRIAL The patients were blinded to their group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath group (Experimental): A conventional physiotherapy program was applied to this group. Additionally, Bobath treatment approach was applied for 10 repetitions during a 30-min session in the experimental group, in addition to the conventional physiotherapy program.
  Interventions: Procedure: Bobath treatment approach; Procedure: Conventional physiotherapy
- Conventional physiotherapy group (Active Comparator): Only conventional physiotherapy program was applied to this group.
  Interventions: Procedure: Conventional physiotherapy

INTERVENTIONS:
Procedure: Bobath treatment approach — scapulothoracic mobilization exercise, reaching in different directions in the supine position and upper extremity weight transfer exercise.
  Other Names: Neurodevelopmental treatment
  Arms: Bobath group
Procedure: Conventional physiotherapy — range of motion, stretching, strengthening exercises, electrotherapy, thermotherapy, balance and mobility exercises and exercises for daily living activities.

SUMMARY:
In this study, it is investigated that whether Bobath approach is superior to conventional physiotherapy in terms of improving hemiplegic shoulder pain, spasticity and upper extremity functionality in stroke patients.

DETAILED DESCRIPTION:
Objective: This study aims to determine the effect of Bobath approach on hemiplegic shoulder pain, spasticity and upper extremity functionality in stroke patients.

Patients and Methods: For this prospective, randomized, controlled and single-blind trial, 30 stroke patients aged 40-65 years with hemiplegic shoulder pain were included. Patients were divided into two groups and randomized into these groups. Only conventional physiotherapy was applied to the control group, whereas both conventional physiotherapy and Bobath exercises were also applied to the experimental group. Visual analog scale (horizontal) for shoulder pain, modified Ashworth scale for spasticity and Fugl-Meyer assessment of the upper extremity for functionality were used for both pre-test and post-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 40 and 65
* Patients who had a stroke for the first time and had a disease duration of at least four weeks
* Patients who were diagnosed with ischemic or hemorrhagic stroke
* Patients who had Brunnstrom stage 3, 4 or 5 and had hemiplegic shoulder pain were included in the study.

Exclusion Criteria:

* Patients with severe cognitive impairment who could not understand simple verbal commands
* Those who had severe dysarthria to prevent verbal communication
* Those with unilateral neglect syndrome
* Those with loss of sensation in the upper extremity of the hemiplegic side
* Those with botulinum toxin-A injected to the hemiplegic upper extremity muscles
* Those with previous shoulder-related trauma or pain history
* Those with other accompanying neurological disease were excluded from the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Fugl-Meyer Assessment score at 30 sessions, 6 weeks | First evaluation: immediately before starting the treatment; the last evaluation: at the end of the treatment of 6 weeks
  Upper extremity functionality, min-max: 0-66, "0" indicates no function of upper extremity, "66" indicates the highest functionality of upper extremity as possible.

SECONDARY OUTCOMES:
Change from baseline Visual Analog Scale (horizontal) value at 30 sessions, 6 weeks | First evaluation: immediately before starting the treatment; the last evaluation: at the end of the treatment of 6 weeks
  Hemiplegic shoulder pain, 0-10 cm scale, "0" shows no pain at hemiplegic shoulder, "10" shows unbearable pain intensity at hemiplegic shoulder
Change from baseline modified Ashworth scale value at 30 sessions, 6 weeks | First evaluation: immediately before starting the treatment; the last evaluation: at the end of the treatment of 6 weeks
  Upper extremity spasticity, 0: No increase in tone, 1: slight increase in tone giving a catch when slight increase in muscle tone manifested by the limb was moved in flexion or extension.
  1+: slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM )
  2: more marked increase in tone but more marked increased in muscle tone through most limb easily flexed
  3: considerable increase in tone, passive movement difficult
  4: limb rigid in flexion or extension

OTHER OUTCOMES:
Change from baseline Brunnstrom Motor Recovery Staging value at 30 sessions, 6 weeks | First evaluation: immediately before starting the treatment; the last evaluation: at the end of the treatment of 6 weeks
  Upper extremity motor evaluation,

CONTACTS AND LOCATIONS:
Overall Officials: NAZLI GÜNGÖR, PT,MSc, Principal Investigator — Istanbul Arel University
Locations (1):
- University of Health Sciences, Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huseyinsinoglu BE, Ozdincler AR, Krespi Y. Bobath Concept versus constraint-induced movement therapy to improve arm functional recovery in stroke patients: a randomized controlled trial. Clin Rehabil. 2012 Aug;26(8):705-15. doi: 10.1177/0269215511431903. Epub 2012 Jan 18. PMID 22257503
- [Background] Tang QP, Yang QD, Wu YH, Wang GQ, Huang ZL, Liu ZJ, Huang XS, Zhou L, Yang PM, Fan ZY. Effects of problem-oriented willed-movement therapy on motor abilities for people with poststroke cognitive deficits. Phys Ther. 2005 Oct;85(10):1020-33. PMID 16180951
- [Background] Langhammer B, Stanghelle JK. Bobath or motor relearning programme? A comparison of two different approaches of physiotherapy in stroke rehabilitation: a randomized controlled study. Clin Rehabil. 2000 Aug;14(4):361-9. doi: 10.1191/0269215500cr338oa. PMID 10945420
- [Background] Suputtitada A, Suwanwela NC, Tumvitee S. Effectiveness of constraint-induced movement therapy in chronic stroke patients. J Med Assoc Thai. 2004 Dec;87(12):1482-90. PMID 15822545
- [Background] Platz T, Eickhof C, van Kaick S, Engel U, Pinkowski C, Kalok S, Pause M. Impairment-oriented training or Bobath therapy for severe arm paresis after stroke: a single-blind, multicentre randomized controlled trial. Clin Rehabil. 2005 Oct;19(7):714-24. doi: 10.1191/0269215505cr904oa. PMID 16250190
- [Background] Hafsteinsdottir TB, Kappelle J, Grypdonck MH, Algra A. Effects of Bobath-based therapy on depression, shoulder pain and health-related quality of life in patients after stroke. J Rehabil Med. 2007 Oct;39(8):627-32. doi: 10.2340/16501977-0097. PMID 17896054
- [Background] Fazekas G, Horvath M, Troznai T, Toth A. Robot-mediated upper limb physiotherapy for patients with spastic hemiparesis: a preliminary study. J Rehabil Med. 2007 Sep;39(7):580-2. doi: 10.2340/16501977-0087. PMID 17724559
- [Background] van Vliet PM, Lincoln NB, Foxall A. Comparison of Bobath based and movement science based treatment for stroke: a randomised controlled trial. J Neurol Neurosurg Psychiatry. 2005 Apr;76(4):503-8. doi: 10.1136/jnnp.2004.040436. PMID 15774435
- [Background] van der Lee JH, Wagenaar RC, Lankhorst GJ, Vogelaar TW, Deville WL, Bouter LM. Forced use of the upper extremity in chronic stroke patients: results from a single-blind randomized clinical trial. Stroke. 1999 Nov;30(11):2369-75. doi: 10.1161/01.str.30.11.2369. PMID 10548673
- [Background] Arya KN, Verma R, Garg RK, Sharma VP, Agarwal M, Aggarwal GG. Meaningful task-specific training (MTST) for stroke rehabilitation: a randomized controlled trial. Top Stroke Rehabil. 2012 May-Jun;19(3):193-211. doi: 10.1310/tsr1903-193. PMID 22668675
- [Background] Wang RY, Chen HI, Chen CY, Yang YR. Efficacy of Bobath versus orthopaedic approach on impairment and function at different motor recovery stages after stroke: a randomized controlled study. Clin Rehabil. 2005 Mar;19(2):155-64. doi: 10.1191/0269215505cr850oa. PMID 15759530